CLINICAL TRIAL: NCT03498144
Title: Evaluation of Acquired Punctal Stenosis by Using Anterior Segment Optical Coherence Tomography (AS-OCT)
Brief Title: Diagnosis of Acquired Punctal Stenosis Using Anterior Segment Optical Coherence Tomography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Heba Radi AttaAllah, Lecturer of Ophthalmology/ Ophthalmology department/Faculty of Medicine/(Principal Investigator), Minia University
Other Study IDs: 62-2/2018
Record Dates: First submitted 2018-04-02; First posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Punctal Stenosis
Keywords: acquired punctal stenosis; epiphora; lower punctum; AS-OCT
MeSH Terms: conditions — Lacrimal Apparatus Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with acquired punctal stenosis: Patients with acquired punctal stenosis with epiphora
  Interventions: Device: Anterior segment OCT
- Control subjects: normal subjects, without evidence of any punctal abnormalities.
  Interventions: Device: Anterior segment OCT

INTERVENTIONS:
Device: Anterior segment OCT — lower punctum examination by AS-OCT
  Other Names: (RTVue model-RT100, with cornea/anterior module lens (CAM system )

SUMMARY:
Purpose of the study

To evaluate the lower puntum dimensions in cases of acquired punctal stenosis(APS), using anterior segment optical coherence tomography (AS-OCT).

DETAILED DESCRIPTION:
(B)Examination:

1. External examination: should be done to rule out causes of watering other than punctal stenosis (facial palsy, lacrimal pump failure, swelling in lacrimal sac area and regurge test)
2. Slit lamp examination: for tear meniscus, lid margin, conjunctiva and punctual orifice
3. Fluorescein dye disappearance test: performed with a drop of 2% fluorescein in lower conjunctival sac, patient is instructed not to wipe the eyes. After 5 minutes, presence of staining in the tear film is assessed with cobalt blue filter.
4. Probing and lacrimal syringing, if patent confirms punctal stenosis to be the cause of epiphora rather than block in the lower lacrimal drainage system.
5. Anterior segment optical coherence tomography examination (AS-OCT) for the lower punctum: measuring the outer puntcal diametre, inner punctal diameter and punctal depth.

Examination of the lower punctum was performed using Spectral Domain OCT machine; RTVue model-RT100 CAM system (Optovue Inc., Fremont, CA, USA) version 6.2, by attaching the cornea/anterior module lens (CAM). CAM lens has a wide-angle, high-magnification lens of 10 mm working distance. The axial resolution was 5 μm, and the lateral resolution was 8 μm. The scan beam has wavelength of 840 ± 10 nm. The two red external illumination (light emitting diode ) LED on headrest were approximated on each side of the lower punctum for proper illumination and imaging of the punctum. Gentle eversion of the medial part of the lower lid was performed to expose the lower lid punctum, so the vertical canaliculus was brought to be at an axial plain without undue stretching or pressure to the lower lid. Line scan was the used examination scan, containing 1020 A-scans/line, and is 8mm in length.

Measurements of the external punctal diameter, internal punctal diameter, and punctal depth were performed on the B-scan image of the lower punctum (by selecting it from the Review window), using distance measurement tool. External punctal diameter was measured as a line connecting highest points on the medial and lateral punctal walls. Internal punctal diameter was measured as a horizontal line just above the narrowing. The distance between the line representing the external punctal diameter and the floor of the punctum was calculated and referred to the punctal depth

Results:

Data wil be collected and statistically analysed

ELIGIBILITY:
Inclusion Criteria:

Patients with acquired punctal stenosis

Exclusion Criteria:

1. Punctal agenesis
2. Congenital punctal stenosis
3. Allergic occlusion
4. Lid malposition
5. Canalicular, nasolacrimal, sac and duct obstruction
6. Previous eyelid or lacrimal drainage surgery
7. Untreated conjunctivitis, blepharitis

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults with acquired punctal stenosis
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Lower punctum dimensions in cases with acquired punctual stenosis, compared with lower punctal dimensions in normal subjects | one month
  External punctum diameter measured in µm, internal punctum diameter, measured in µ m, punctal depth measured in µ m

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soiberman U, Kakizaki H, Selva D, Leibovitch I. Punctal stenosis: definition, diagnosis, and treatment. Clin Ophthalmol. 2012;6:1011-8. doi: 10.2147/OPTH.S31904. Epub 2012 Jul 3. PMID 22848141
- [Background] Kakizaki H, Takahashi Y, Iwaki M, Nakano T, Asamoto K, Ikeda H, Goto E, Selva D, Leibovitch I. Punctal and canalicular anatomy: implications for canalicular occlusion in severe dry eye. Am J Ophthalmol. 2012 Feb;153(2):229-237.e1. doi: 10.1016/j.ajo.2011.07.010. Epub 2011 Oct 6. PMID 21982102
- [Background] Kashkouli MB, Pakdel F, Kiavash V. Assessment and management of proximal and incomplete symptomatic obstruction of the lacrimal drainage system. Middle East Afr J Ophthalmol. 2012 Jan;19(1):60-9. doi: 10.4103/0974-9233.92117. PMID 22346116
- [Background] Wawrzynski JR, Smith J, Sharma A, Saleh GM. Optical coherence tomography imaging of the proximal lacrimal system. Orbit. 2014 Dec;33(6):428-32. doi: 10.3109/01676830.2014.949793. Epub 2014 Sep 12. PMID 25215411